CLINICAL TRIAL: NCT06764056
Title: Characterization and Management of Metabolic Dysfunction-Associated Fatty Liver Disease (MAFLD) Through an Individualized Nutritionnal Approach and Semaglutide Therapy.
Brief Title: Characterization and Management of Metabolic Dysfunction-Associated Fatty Liver Disease (MAFLD)
Acronym: METAfoie
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Responsible Party: Principal Investigator, Fannie Lajeunesse-Trempe, Principal Investigator, Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-4271
Record Dates: First submitted 2024-12-18; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Metabolic Associated Fatty Liver Disease; Metabolic Associated-dysfunction Steatohepatitis (MASH); Obesity
Keywords: Obesity; Metabolic associated fatty liver disease; GLP-1 receptor analogs; Pharmacotherapy; Nutrition; Transient elastography; Semaglutide; Microbiome; Lipidomics
MeSH Terms: conditions — Obesity | interventions — semaglutide; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nutrition (Active Comparator): This arm will only participate in an individualized nutritionnal approach.
  Interventions: Other: Diet
- Nutrition + Semaglutide (Active Comparator): This arm will initiate a pharmacological intervention to treat obesity (Semaglutide) and will participate in an individualized nutritionnal approach.
  Interventions: Drug: semaglutide; Other: Diet
- Semaglutide (Active Comparator): This arm will only initiate a pharmacological intervention to treat obesity (Semaglutide)
  Interventions: Drug: semaglutide

INTERVENTIONS:
Drug: semaglutide — Participants receiving this intervention will be starting with a dose of semaglutide 0.25 mg. Physicians will follow Wegovy® Dosing Schedule guidelines, ending with a final dose of 2.4 mg at the fifth month. Type 2 diabetes participants wishing to stop at 1.0 mg will be allowed.
  Arms: Nutrition + Semaglutide; Semaglutide
Other: Diet — Participants receiving this intervention will be seeing a registered dietician at each visit. The individualized approach will be based on recent literature (mostly hypocaloric) by using different methods.
  Other Names: Individualized nutritionnal intervention; Nutritionnal counselling
  Arms: Nutrition; Nutrition + Semaglutide

SUMMARY:
The goal of this clinical trial is to improve the treatment of hepatic steatosis associated with obesity with pharmacological and nutritionnal approaches. The main question it aims to answer is:

Does an individualized nutritionnal approach with a dietician combined with medication targeting obesity is the most efficient way to treat hepatic steatosis associated with obesity?

Participants will either participate in one of three groups:

* Nutrition: Participant will only have a regular follow-up with a registered dietician;
* Nutrition + Semaglutide: Participants will start a new medication targeting obesity and will have a regular follow-up with a registered dietician;
* Semaglutide: Participants will start a new medication targeting obesity.

DETAILED DESCRIPTION:
Participants in each group will be followed during a year for 4 timepoints (0, 3, 6 and 12 months). Blood and feces samples, anthropometric measures, transient elastography measurements and health questionnaires will be assessed at each timepoint.

The nutritionnal intervention targeting hepatic steastosis associated with obesity will use conclusions from a systematic review we conducted on nutritionnal approaches to treat liver steatosis.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 30 and 50 kg/m2;
* Stade 2 or 3 (S2 or S3) hepatic steatosis with or without liver fibrosis.

Exclusion Criteria:

* Type 1 diabetes diagnosis;
* Alcohol consumption exceeding recommendations [>140 g/week (women) and >210 g/week (men)];
* Known chronic hepatic disease non-steatotic at the entry of the study (Wilson's disease, hemochromatosis, alpha-1-antitrypsin deficiency, viral hepatitis, auto-immune hepatitis, etc.);
* Pharmacological treatment targeting obesity active or ended in the last 3 months;
* Bariatric surgery;
* Gastro-intestinal pathologies (GI cancers, IBD, etc.);
* Capsulated probiotics consumption;
* Antibiotic treatment in the last 3 months;
* Pregnancy;
* Cirrhosis diagnosis (hepatic decompensation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Liver Steatosis | From enrollment to the end of the clinical trial at 12 months (for 4 visits)
  Transient elastography is an ultrasound-based modality that is non-invasive and measures the degree of steatosis with the controlled attenuation parameter (CAP; dB/m) and liver stiffness (kPa).This method will be used at each visit to follow the progression and the efficiency of the interventions.
  The following ranges will be use to classify hepatic steatosis based on CAP (dB/m) (specific to FibroScan®): S0 (< 302), S1 (302-331), S2 (331-337) and S3 (>337).
Liver Stiffness | From enrollment to the end of the clinical trial at 12 months (for 4 visits)
  Transient elastography is an ultrasound-based modality that is non-invasive and measures the degree of steatosis with the controlled attenuation parameter (CAP; dB/m) and liver stiffness (kPa).This method will be used at each visit to follow the progression and the efficiency of the interventions.
  The following ranges will be use to classify hepatic fibrosis based on liver stiffness (kPa) (specific to FibroScan®): F0-F1 (< 8.0), F2 (8.9-9.7), F3 (9.7-13.6) and F4 (>13.6).

SECONDARY OUTCOMES:
Liver function (biochemistry) | From enrollment to the end of the clinical trial at 12 months (for 4 visits)
  Blood samples will be drawn at each visit to assess the following measures:
  liver enzymes (aspartate aminotransferase [AST], alanine aminotransferase [ALT], gamma-glutamyl transferase [GGT], alkaline phosphatase [ALP]), total bilirubin and albumin. Liver scores will also be calculated: fatty liver index (FLI) and fibrosis-4 index (FIB-4)
  The following normal ranges will be used:
  * AST : [8-33] U/L;
  * ALT : [10-40] U/L;
  * GGT : [2-30] U/L;
  * ALP : [30-120] U/L;
  * Total bilirubin : [5-21] umol/L;
  * Albumin : [35-30] g/L.
  * FLI : <30 : Low risk of hepatic steatosis ; >60 : High risk of hepatic steatosis.
  * FIB-4 : >3.48 : High risk of cirrhosis
Lipid panel | From enrollment to the end of the clinical trial at 12 months (for 4 visits)
  Blood samples will be drawn at each visit to assess the lipid panel.
  The following ranges will be used:
  * triglycerides: < 1.5 mmol/L;
  * total cholesterol: < 5.20 mmol/L;
  * LDL-cholesterol: < 2.59 mmol/L;
  * HDL-cholesterol: > 1.55 mmol/L;
Change from Baseline in the gut microbiota diversity | From enrollment to the end of the clinical trial at 12 months (for 4 visits)
  The composition of the gut microbiota will be measured at each visit with the participants' stool samples. The difference between the concentration of gut microbiota diversity (bacteria, families, phyllum, etc.) will be analyzed.
Change from Baseline in blood lipids and metabolites | From enrollment to the end of the clinical trial at 12 months (for 4 visits)
  We will perform lipidomic and metabolomic measures with blood samples of each visit with liquid chromatography coupled with mass spectrometry (LC-MS/MS).
Glucose | From enrollment to the end of the clinical trial at 12 months (for 4 visits)
  Blood samples will be drawn at each visit to assess the glucose.
  The following range will be used:
  - glucose: < 5.6 mmol/L;
Insulin | From enrollment to the end of the clinical trial at 12 months (for 4 visits)
  Blood samples will be drawn at each visit to assess insulin
  The following range will be used:
  - insuline: [20-60] pmol/L;
Glycated hemoglobin | From enrollment to the end of the clinical trial at 12 months (for 4 visits)
  Blood samples will be drawn at each visit to assess HbA1c
  The following range will be used:
  - HbA1c: < 6.5 %;
C-reactive protein | From enrollment to the end of the clinical trial at 12 months (for 4 visits)
  Blood samples will be drawn at each visit to assess the c-reactive protein
  The following range will be used:
  - CRP: < 10 mg/L.
Liver enzymes | From enrollment to the end of the clinical trial at 12 months (for 4 visits)
  Blood samples will be drawn at each visit to assess the following measures:
  liver enzymes (aspartate aminotransferase [AST], alanine aminotransferase [ALT], gamma-glutamyl transferase [GGT] and alkaline phosphatase [ALP]),
  The following normal ranges will be used:
  * AST : [8-33] U/L;
  * ALT : [10-40] U/L;
  * GGT : [2-30] U/L;
  * ALP : [30-120] U/L.
Fatty liver index (FLI) | From enrollment to the end of the clinical trial at 12 months (for 4 visits)
  The Fatty liver index (FLI) is a non-invasive score to calculate liver steatosis (using BMI, WC, TG and GGT).
  The following ranges will be used:
  * <30 : Low risk of hepatic steatosis ;
  * >60 : High risk of hepatic steatosis.
Fibrosis-4 index (FIB-4) | From enrollment to the end of the clinical trial at 12 months (for 4 visits)
  The fibrosis-4 index (FIB-4) is a non-invasive score to calculate liver fibrosis (using Age, AST, ALT and Platelet count).
  The following normal range will be used:
  - <30 : Low risk of hepatic steatosis ; >60 : High risk of hepatic steatosis. fatty liver index (FLI) and
  The following range will be used:
  - FIB-4 : >3.48 : High risk of cirrhosis

CONTACTS AND LOCATIONS:
Overall Officials: Fannie Lajeunesse-Trempe, MD., Ph.D., Principal Investigator — Centre de recherche de l'Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval
Locations (1):
- Centre de recherche de l'Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No